CLINICAL TRIAL: NCT00016835
Title: Treating Periodontal Infection: Effects on Glycemic Control in People With Type 2 Diabetes
Brief Title: Treating Periodontal Infection: Effects on Glycemic
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, George W. Taylor, Professor Emeritus, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDCR-03; 5R01DE013796-03 (NIH)
Record Dates: First submitted 2001-06-05; First posted 2001-06-07 (Estimated); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Periodontal Disease; Diabetes Mellitus, Type 2
Keywords: Type 2 diabetes mellitus; Glycemic control; Periodontal therapy
MeSH Terms: conditions — Periodontal Diseases; Diabetes Mellitus, Type 2 | interventions — Dental Scaling; Metronidazole; Doxycycline

STUDY DESIGN:
Intervention Model Description: Study participants were randomized into 3 groups for the initial non-surgical treatment appointment. One group received supra-gingival scaling and placebo, one group received non-surgical periodontal supra- and sub-gingival scaling plus metronidazole and one group received non-surgical periodontal supra- and sub-gingival scaling plus doxycycline. All three groups received 3-month follow-up visits for 15 months and the group receiving supra-gingival scaling and placebo at the initial visit received supra- and sub-gingival scaling at the 9-month follow-up visit.
Who Masked: Participant, Care Provider
Masking Description: Participants and examiners were unaware of the type of medication and examiners were also unaware of the type of periodontal therapy the participants receive
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supra-gingival scaling and placebo (Active Comparator): This group receives a placebo (instead of systemic antibiotic), supra-gingival oral prophylaxis, and ultrasonic removal of supra-gingival calculus with water irrigation at the initial treatment visit. At the 9-month follow-up visit, this group will receive sub-gingival ultrasonic scaling with povidone-iodine irrigation.
  This group also receives regular follow-up evaluations and site-specific mechanical periodontal therapy, at 3-month intervals, for approximately 15 months.
  Interventions: Procedure: Supra-gingival scaling and placebo
- Subgingival scaling and metronidazole (Experimental): This group receives ultrasonic scaling with local anesthesia (as needed), local antimicrobial treatment with povidone-iodine irrigation, and metronidazole as an oral systemic antibiotic at the initial treatment visit.
  This group also receives regular follow-up evaluations and site-specific mechanical periodontal therapy, at 3-month intervals, for approximately 15 months.
  Interventions: Procedure: Subgingival scaling and metronidazole
- Subgingival scaling and doxycycline (Experimental): This group receives ultrasonic scaling with local anesthesia (as needed), local antimicrobial treatment with povidone-iodine irrigation, and doxycycline as an oral systemic antibiotic at the initial treatment visit.
  This group also receives regular follow-up evaluations and site-specific mechanical periodontal therapy, at 3-month intervals, for approximately 15 months.
  Interventions: Procedure: Subgingival scaling and doxycycline

INTERVENTIONS:
Procedure: Supra-gingival scaling and placebo — Included in arm/group description.
  Arms: Supra-gingival scaling and placebo
Procedure: Subgingival scaling and metronidazole — Included in arm/group description.
  Arms: Subgingival scaling and metronidazole
Procedure: Subgingival scaling and doxycycline — Included in arm/group description.
  Arms: Subgingival scaling and doxycycline

SUMMARY:
The purpose of this project is to obtain important preliminary data necessary to support design of a full scale, multicenter randomized clinical trial (RCT) to evaluate the effect of treating periodontal infection on glycemic control in type 2 diabetes mellitus.

DETAILED DESCRIPTION:
There is compelling epidemiological and clinical evidence to suggest that periodontal infection adversely affects glycemic control in people with type 2 diabetes mellitus. The purpose of this pilot project is to obtain important preliminary data necessary to support design of a full scale, multi-center randomized clinical trial (RCT) to evaluate the effect of treating periodontal infection on glycemic control in individuals with type 2 diabetes mellitus. This current project involves treating periodontal infection to obtain estimates of changes and the variability of those changes over time in the established primary endpoint, hemoglobin A1c (HbA1c). This project will also explore use of several potential secondary endpoints including levels of periodontitis and glucose metabolism-related inflammatory mediators (TNF-alpha, IL-1-beta, IL-6), serum cholesterol, triglyceride and lipids. Subjects are randomly assigned to 1 of three possible groups for comprehensive periodontal examination, specimen collection, mechanical periodontal therapy and oral systemic antibiotics or placebo, and regular follow-up evaluations and site-specific mechanical periodontal therapy, at 3-month intervals, for approximately 15 months. Two groups receive ultrasonic scaling with local anesthesia (as needed), local antimicrobial treatment with povidone-iodine irrigation, and an oral systemic antibiotic (either doxycycline or metronidazole) at the initial treatment visit. The third group ("controls") receives a placebo and supra-gingival oral prophylaxis and ultrasonic removal of supra-gingival calculus with water irrigation at the initial treatment visit. At the 9-month follow-up visit, "controls" receive sub-gingival ultrasonic scaling with povidone-iodine irrigation.

Results from this pilot project will be used as preliminary data to support design of an immediate follow-up proposal to NIH/NIDCR for funding a multi-center RCT to evaluate the effect of treating periodontal infection on glycemic control in type 2 diabetes. If results from the full scale clinical trial provide evidence that treating periodontal infection contributes to improved glycemic control, then diagnosis and treatment of periodontal infection in subjects with type 2 diabetes could be substantiated as an important component in management of diabetes.

ELIGIBILITY:
Inclusion Criteria

* Subjects must be 18 years of age or older,
* have at least six natural teeth,
* have established periodontal disease (established at the screening examination),
* have a history of type 2 diabetes of at least six months with HbAlc > 7.1%.

Exclusion Criteria

* Subjects will be excluded from the study if they are presently under the care of a periodontist;
* have had antibiotic treatment within the previous three months;
* have conditions that require antibiotic prophylaxis for dental treatment;
* have allergies to iodine, doxycycline, metronidazole, or chlorhexidine;
* have blood dyscrasias;
* are pregnant or breast feeding;
* have severe cognitive or communication impairment;
* have a cardiac pacemaker;
* are under cancer chemotherapy;
* are medically unstable or have a life expectancy of less than two years;
* are currently taking disulfiram, phenobarbital, lithium, terfenadine, astemizole, or warfarin;
* or are out of town or otherwise unavailable for more than three consecutive months of the year.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2001-10-17 (Actual); Primary Completion 2004-09-03 (Actual); Study Completion 2004-09-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George W. Taylor, DMD, Dr.PH, Principal Investigator — University of Michigan
Locations (1):
- Department of Cariology, Restorative Sciences and Endodontics, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
There is no current plan to share data with other researchers at this time